CLINICAL TRIAL: NCT03128853
Title: Spot-Check Noninvasive Hemoglobin (SpHb) Repeatability and Reproducibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-18216
Record Dates: First submitted 2017-04-14; First posted 2017-04-25 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Anemia; Healthy
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test subjects (Experimental): Each subject receives the Rad-67 and DCI Mini sensor that will measure hemoglobin repeatedly in order to compare those measurements against a blood sample reference.
  Interventions: Device: Rad-67 and DCI Mini Sensor

INTERVENTIONS:
Device: Rad-67 and DCI Mini Sensor

SUMMARY:
Single-arm study to investigate the repeatability and reproducibility of SpHb measurements from the Rad-67 and DCI Mini sensor.

DETAILED DESCRIPTION:
This study aims to evaluate the repeatability and reproducibility of Masimo's pulse CO-Oximeter and sensor to determine the device and sensor's precision in SpHb measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age one month and older
* Weight greater than or equal to 3 kg
* The subject or the subject's legally authorized representative has given written informed consent/assent to participate in the study

Exclusion Criteria:

* Decision-impaired adult and pediatric patients who are unable to give informed consent/assent
* Decision-impaired adult on behalf of a pediatric patient who is unable to assent
* Subjects with skin abnormalities at the planned application sites that may interfere with sensor application, per directions-for-use (DFU) or trans-illumination of the site, such as burns, scar tissue, nail polish, acrylic nails, infections, abnormalities, etc.
* Subjects deemed not suitable for the study at the discretion of the investigator
* Subjects unlikely to be able to refrain from excessive motion during data collection. Excessive motion includes postural changes, making hand gestures, involuntary muscular movements, etc.

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Repeatability and reproducibility of CO-oximeter and sensor | 120 minutes
  The Repeatability and Reproducibility of the sensor will be assessed by varying the testing conditions (operator/device, finger, subject, and repetition) to determine the device and sensor's precision in SpHb measurements.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Masimo Clinical Laboratory, Irvine, California
  - Site 1, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No